CLINICAL TRIAL: NCT01518374
Title: Clinical Evaluation of Florbetapir F 18 (18F-AV-45)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A14
Record Dates: First submitted 2011-07-20; First posted 2012-01-26 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Neurodegenerative Diseases
Keywords: Male or female subjects at least 18 years of age; AD; MCI
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neurodegenerative Diseases | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Florbetapir-PET Scans (Experimental)
  Interventions: Drug: Florbetapir F 18

INTERVENTIONS:
Drug: Florbetapir F 18 — 370 MBq (10 mCi)
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This protocol is designed to standardize imaging studies using florbetapir F 18 PET to provide information on amyloid burden in subjects participating in other studies (companion protocol) such as longitudinal studies of aging and studies of biomarkers for neurodegenerative diseases.

ELIGIBILITY:
Subjects who meet all of the following criteria are eligible to enroll in this study:

1. Male or female subjects at least 18 years of age;
2. Subjects who sign an IRB approved informed consent prior to any study procedures. Where subjects are deemed incapable of informed consent, a legally authorized representative may provide consent, with the subject's documented assent; and
3. Subjects who in the opinion of the investigator can tolerate the PET scan procedures.

Subjects will be excluded from enrollment if they:

1. Have clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances as indicated by history, which in the opinion of the investigator might pose a potential safety risk to the subject;
2. Have current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following:

   * cardiac surgery or myocardial infarction within the last 4 weeks;
   * unstable angina;
   * acute decompensated congestive heart failure or class IV heart failure;
   * current significant cardiac arrhythmia or conduction disturbance, particularly those resulting in ventricular fibrillation, or causing syncope, or near syncope;
   * uncontrolled high blood pressure; or
   * QTc > 450 msec (by history or for patients with cardiac disease by screening evaluation in companion study)

   Before enrolling a patient with any of the above conditions, the investigator must have performed a cardiac evaluation and obtain permission from the sponsor.
3. Have a history of drug or alcohol abuse within the last year, or prior prolonged history of abuse;
4. Women of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception. Women of childbearing potential must not be pregnant (negative urine beta-hCG at the time of screening and negative urine beta-hCG on the day of imaging) or breastfeeding at screening. Women must avoid becoming pregnant, and must agree to refrain from sexual activity or to use reliable contraceptive methods for 24 hours following administration of Florbetapir F 18 Injection ( such as oral contraceptives for at least three months or an IUD for at least two months prior to the start of the screening visit, or various barrier methods, e.g., diaphragm or combination condom and spermicide);
5. Have a history of relevant severe drug allergy or hypersensitivity (Relevant severe drug allergies should be determined by the PI, and any questions about a subject's eligibility can be directed to Avid. If a subject has a history of severe drug allergies, it may be dangerous for them to participate in a study);
6. Are patients who have received an investigational medication under an FDA IND protocol within the last 30 days. Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication. Patients who have ever participated in an experimental study with an amyloid targeting therapy (e.g., immunotherapy, secretase inhibitor) may not be enrolled without prior sponsor approval unless it can be demonstrated that the patient received only placebo in the course of the trial;
7. Are patients with current clinically significant unstable medical comorbidities, as indicated by history or physical exam, that pose a potential safety risk to the subject.
8. Are patients who have received a radiopharmaceutical for imaging or therapy within the past 24 hours prior to the imaging session for this study. If another radiotracer is required in the companion protocol, patients may be able to receive a radiopharmaceutical for imaging or therapy within the 24 hours prior to the imaging session with prior sponsor approval and at the discretion of the investigator.; and
9. Are patients who, in the opinion of the investigator, are otherwise unsuitable for a study of this type.

If at the time of enrollment subjects do not meet all eligibility criteria, the subjects may still be enrolled if documentation is provided demonstrating that the subject will meet all criteria at the time of the first imaging procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1768 (Actual)
Dates: Start 2009-12; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (24):
- United States (24):
  - Banner Health, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - UC Davis, Davis, California
  - UC Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - UC Irvine, Orange, California
  - UC San Francisco, San Francisco, California
  - UC San Francisco Memory Center, San Francisco, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mt. Sinai Medical Center, Miami Beach, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Jefferson, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - University of Tennessee, Knoxville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - UTSW, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All enrolled subjects who received an injection of florbetapir and completed safety assessment were considered to have completed the study.
Pre-assignment Details: This was a standardized imaging protocol designed to support companion studies where amyloid imaging was used as a biomarker in longitudinal studies of aging or studies of biomarkers for neurodegenerative diseases. Subjects had to meet additional inclusion/exclusion criteria for the companion protocol before being injected and imaged under A14.
Period: Overall Study
Arm/Group | Florbetapir-PET Scans
Started | 1768
Completed | 1761
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Florbetapir-PET Scans
Number analyzed (Participants) | 1768
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 6 participants did not have baseline age in the database
  years
    number analyzed (Participants) | 1762
    (all) | 68.3 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 920
  Male | 848
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 233
  White | 1487
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1768

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events Considered Related to Florbetapir Administration
Description: Frequency of treatment-emergent adverse events considered related to florbetapir administration by the study investigator. Related events with a frequency > 0.2% are reported.
  (note: all treatment-emergent adverse events, regardless of relatedness designation, are reported in "Adverse Events" section below)
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Florbetapir-PET Scans
Number analyzed (Participants) | 1768
Participants
  Headache | 21
  Injection site pain | 6
  Dizziness | 5
  Nausea | 5
  Fatigue | 4
  Back pain | 4
  Dry mouth | 4

ADVERSE EVENTS:
Time Frame: Within 48 hours of florbetapir injection
Description: Note: adverse events results differ from results reported above because this section reports ALL adverse events, regardless of relatedness designation by the investigator.
Arm/Group | Florbetapir-PET Scans
All-Cause Mortality (participants affected / at risk) | 0/1768
Serious Adverse Events (participants affected / at risk) | 1/1768
Other Adverse Events (participants affected / at risk) | 111/1768
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Florbetapir-PET Scans (N=1768)
Ischaemic stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Florbetapir-PET Scans (N=1768)
Headache (Nervous system disorders) | 47
Nausea (Gastrointestinal disorders) | 14
Fatigue (General disorders) | 12
Dizziness (Nervous system disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 11
Injection site pain (General disorders) | 8
Dry mouth (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2013-02-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT01518374/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT01518374/SAP_001.pdf